CLINICAL TRIAL: NCT06258330
Title: A Phase I, Open-Label Multicenter Study of AM003 Dose Escalation, Administered Intratumorally to Patients With Locally Advanced and Metastatic Solid Tumors
Brief Title: Study of AM003 in Patients With Locally Advanced and Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aummune Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AM003-FIH-001
Record Dates: First submitted 2022-06-01; First posted 2024-02-14 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor
Keywords: Phase 1; Dose escalation; Personalized treatment

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 - low dose (Experimental): AM003 34 mg
  Interventions: Drug: AM003
- Cohort 2 - mid dose (Experimental): AM003 68 mg
  Interventions: Drug: AM003
- Cohort 3 - high dose (Experimental): AM003 136 mg
  Interventions: Drug: AM003

INTERVENTIONS:
Drug: AM003 — Bispecific Personalized Aptamer for intratumoral administration

SUMMARY:
This is a phase 1, first-in-human study to assess the safety and tolerability of AM003 in patients with locally advanced and metastatic solid tumors

DETAILED DESCRIPTION:
This is a phase 1, open-label , multicenter dose escalation trial evaluating the safety and tolerability of AM003 , administered intratumorally to patients with locally advanced and metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent.
2. Capable of providing signed informed consent, which includes compliance with the requirements of this protocol.
3. Participants with histologically confirmed locally advanced/metastatic solid tumors who received and progressed after or were intolerant to at least 1 prior systemic therapy (unless no Standard of Care therapy exists) and are not candidates for any therapy known to confer clinical benefit.

   Eligible for recruitment are participants with a variety of solid tumors such as:
   * Head and neck cancers
   * Thyroid cancers
   * Soft tissue sarcoma
   * Colorectal cancers
   * Skin (melanoma and non-melanoma),
   * other cancer indications may be considered, but require sponsor approval NOTE: prior exposure to PD-1 or PDL-1 inhibitors are permitted.
4. Lesions that are amenable to IT injection (by visual inspection, palpation, ultrasound or CT guidance). At least one measurable lesion must be amenable to both IT injection and biopsy. A measurable distant, discrete lesion that is also amenable to biopsy is optional.
5. All participants must have measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam, in at least one dimension (longest diameter to be recorded).

   5.1. For cohort 1 (dose level 1) participant must have at least one lesion ≥ 1.5 cm 5.2. For cohorts 2 and 3 (dose levels 2&3), participant should preferably have at least one lesion ≥ 2.5cm and ≥ 5cm for cohorts 2 and 3 respectively. For cases in which no such single lesion can be identified, the total dose of AM003 may be split among several lesions or between a lesion and local SC administration(s).
6. Personalized AM003 sequence identified for the participant during the pre-screening period or previous related studies.
7. Eastern Cooperative Oncology Group (ECOG) performance status score ≤1.
8. Life expectancy of >3 months.
9. Have adequate organ function as defined by the following laboratory values within 7 days of dosing the first dose of AM003:

   System Lab Value Hematology Absolute neutrophil count ≥ 1,000/μl Platelets ≥ 100,000/ul Hemoglobin ≥ 9 g/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Partial Thromboplastin Time (PTT) or Activated Partial Thromboplastin Time(aPTT) <1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Renal Serum creatinine ≤ 1.5 x ULN or creatinine clearance (observed or estimated using the Cockcroft-Gault equation) ≥ 45 mL/min Hepatic Total bilirubin ≤ 1.5 x ULN (except participants with Gilbert syndrome who must have a total bilirubin level of < 3.0 x ULN) AST/ALT ≤ 3.0 x upper limits of normal (ULN) or ≤ 5.0 x ULN in participants with hepatocellular carcinoma or if liver metastases are present
10. Male and female participants of child-bearing potential must agree to use highly effective contraception while enrolled in the study and receiving the experimental drug, and for at least 3 months after the last treatment. Female participants of child-bearing potential must have a negative serum pregnancy test confirmed within 7 days of receiving the initial dose of AM003 therapy.

Exclusion Criteria:

1. Clinical evidence of active central nervous system (CNS) disease NOTE: Participants are eligible if brain metastases are adequately treated and participants are neurologically stable (except for residual signs or symptoms related to the central nervous system (CNS) treatment) for at least 2 weeks prior to enrollment without the use of corticosteroids or are on a stable or decreasing dose of≤ 10 mg daily prednisone (or equivalent)
2. History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to the first date of study treatment.
3. Participants with congestive heart failure (≥NYHA class 3) or unstable angina pectoris.
4. Active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
6. Prior severe hypersensitivity reaction to treatment with a monoclonal antibody
7. Has not fully recovered from any effects of major surgery, and be free of significant detectable infection. Surgeries that required general anesthesia must be completed at least 2 weeks before first study drug administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study drug administration and participants should be recovered.
8. History of organ transplant.
9. Positive antibody and antigen tests for hepatitis virus B (HBV), hepatitis virus C (HCV) and human immunodeficiency virus (HIV). In the case of positive antibodies and a negative antigen test for hepatitis virus B or negative PCR for hepatitis virus C (representing convalescence) inclusion is permitted.
10. Any Serious illness, uncontrolled inter-current illness, psychiatric illness, active of uncontrolled infection or other medical history, including laboratory results, which, in the opinion of the Investigator, would preclude the participant from adhering to the protocol or would increase the risk associated with study participation or study drug administration or interfere with the interpretation of study results.
11. Participant received other investigational therapy, definitive radiation within 2 weeks, immunotherapy or treatment with anticancer medications within 28 days or at least 5 half-lives prior to the first dose of treatment, whichever is less.
12. Participant is currently not recovered to baseline or CTCAE Grade 1 from the AEs due to cancer therapeutics administered more than 28 days prior to the first dose of treatment except for alopecia and peripheral neuropathy
13. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of SAEs, TEAEs assessed by CTCAE v.5.0 | First 28 days of treatment
Number of TEAEs meeting protocol defined DLT criteria | First 28 days of treatment
  Number and percent of participants experiencing dose-limiting toxicities (DLTs), Grade 3 non-hematological adverse AEs, Grade 4 hematological AEs, and discontinuations of study drug due to AE intolerance.

SECONDARY OUTCOMES:
Number of participants responding to treatment by RESICT 1.1 criteria | Duration of the study, estimated to be 6 months
  Estimating the ORR, Disease Control Rate, CR, PR and SD lasting at least 8 weeks by RECIST 1.1
Number of participants responding to treatment by iRECIST criteria | Duration of the study, estimated to be 6 months
  Estimating the ORR, Disease Control Rate, CR, PR and SD lasting at least 8 weeks by iRECIST.
AM003 PK parameters - Cmax | First 5 weeks of treatment
  Maximum concentration (Cmax)
AM003 PK parameters - AUC | First 5 weeks of treatment
  Area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Irit Carmi Levy, PhD, Study Chair — GM and Chief Scientific Officer Aummune
Locations (5):
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No